CLINICAL TRIAL: NCT04948437
Title: Urinary Exosomal Biomarkers of Thyroglobulin and Galectin-3 for Prognosis and Follow-up in Patients of Well-differentiated Thyroid Cancer
Brief Title: Urinary Exosomal Biomarkers of Thyroglobulin and Galectin-3 for Prognosis and Follow-up in Patients of Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012036RIND
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Thyroid Cancer; Papillary Thyroid Cancer; Follicular Thyroid Cancer
Keywords: Exosome; Urine; Biological marker; Thyroglobulin; Galactin-3
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Now, the investigators carried out a prospective study enrolling patients with thyroid cancer, who had received ablative thyroidectomy and /or radioactive iodine therapy for two more years. The investigators' study already enrolled seventy-three patients with thyroid cancer, and the investigators plan to enroll 30 new patients in this consecutive research study. All patients received total thyroidectomy under clinically surgical judgement in initial therapeutic option. The investigators also further found some difference between papillary thyroid cancer and follicular thyroid cancer, and the investigators will continue annually to closely monitor the change of U-Ex Tg and urinary exosomal galectin-3 between differently cellular types of thyroid cancers.

DETAILED DESCRIPTION:
Although, most thyroid cancers are clinically endocrine tumors of low malignancy, most patients usually receive radioactive iodine-131 treatment and thyroidectomy. Such patients are followed up with thyroid ultrasound and continuous serum thyroglobulin assessment after surgery. Previous studies have shown that one third of well-differentiated thyroid cancers may be transformed into poorly differentiated or even fatal malignant tumors during disease progression, but the efficacy of surgery, chemotherapy and external radiation therapy is not significant. . In other words, effective treatment strategies and tracking models will be very important, including surgical removal of thyroid cancer, radioactive iodine-131 treatment, and tracking of biomarkers in thyroid cancer.

When thyroid cancer cells are poorly differentiated, cell dedifferentiation is a key factor for malignant transformation and invasion. Usually in papillary thyroid carcinoma and follicular thyroid carcinoma, the cancer cells will gradually dedifferentiate, and undifferentiated thyroid carcinoma is the final result. Therefore, the investigators try to find biomarkers and therapeutic tracking targets based on the expression of exosomal proteins in urine. The basis of this clinical study depends on the previous basic experiments of culturing undifferentiated thyroid cancer cells.

Exosomes are nanosomes that are secreted into the extracellular environment. Cancer cell-derived exosomes can be found in the plasma, saliva, urine and other body fluids of cancer patients. The investigators will analyze exosomal proteins in urine, including thyroglobulin and galectin-3, and discover early prognostic biomarkers in urine through the prospectively observation study. The investigators have published preliminary research papers on 16 patients with thyroid mastoid carcinoma and follicular carcinoma in international scientific journals. During the period of surgery and further radioactive iodine-131 therapy, including before and one day after surgery, 3 months and 6 months after surgery, the urinary biomarkers of thyroglobulin and galectin-3 in the urine were analyzed at different stages . A prospective study currently in progress has enrolled 73 patients with thyroid mastoid carcinoma and follicular carcinoma. After thyroidectomy, urine was collected during outpatient follow-up and analyzed for exosome biomarkers in the urine. During the first two years of this project, such new urinary biomarkers of thyroid papillary carcinoma and thyroid follicular carcinoma had shown certain different patterns. The investigators' research team expects to enroll 30 new thyroid cancer patients in this consecutive plan. Under continuous follow-up research, in addition to identifying the clinical application of new biomarker as prognostic predictors for future thyroid cancer patients after surgery, the investigators also plan to observe current patients with thyroid follicular cancer. Up to date, follicular thyroid cancer cannot be diagnosed preoperatively via images or aspiration cytology, because pathology after surgery is the only diagnostic golden rule. According to the observations conducted in the current experiment, the urine exosomal thyroglobulin has the opportunity to be a way to diagnose thyroid follicular carcinoma before surgery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed patients with thyroid papillary, follicular and anaplastic thyroid cancer, post-operation follow up

Exclusion Criteria:

* unclearly diagnosed patients with thyroid papillary, follicular and anaplastic thyroid cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators carried out a prospective study enrolling patients with thyroid cancer, who had received ablative thyroidectomy and /or radioactive iodine therapy for two more years. The study already enrolled seventy-three patients with thyroid cancer, and the investigators plan to enroll 30 new patients in this consecutive research study. All patients received total thyroidectomy under clinically surgical judgement in initial therapeutic option. The investigators also further found some difference between papillary thyroid cancer and follicular thyroid cancer, and we will continue annually to closely monitor the change of U-Ex Tg and urinary exosomal galectin-3 between differently cellular types of thyroid cancers.
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum thyroglobulin level | Within 36 months
  Thyroid function test
Change of serum free T4 level | Within 36 months
  Thyroid function test
Change of serum TSH level | Within 36 months
  Thyroid function test
Change of anti-thyroglobulin level | Within 36 months
  Thyroid function test
Urinary exosomal thyroglobulin detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal galectin-3 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal calprotectin A9 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal transketolase detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal keratin 19 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal angiopoietin-1 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal tissue inhibitor of metalloproteinase detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal keratin 8 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal calprotectin A8 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal annexin II detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal afamin detection | Within 36 months
  Urinary exosomal biomarker

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YUAN WANG, Doctor, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Chih-Yuan Wang, M.D, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No